CLINICAL TRIAL: NCT01900795
Title: A Phase 2a, Single-Center, Randomized, Double-Blind, Double- Dummy, Placebo- and Active-Controlled Analgesic Study of an Oral Dose of V117957 4.5 mg for the Treatment of Postsurgical Pain Due to Third Molar Extraction
Brief Title: An Analgesic Study to of V117957 for the Treatment of Postsurgical Pain Due to Third Molar Extraction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early due to administrative reasons not related to safety.
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OAG2001
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Postsurgical Pain Due to Third Molar Extraction
Keywords: Postsurgical pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- V117957 (Experimental)
  Interventions: Drug: V117957
- Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: V117957 — V117957 4.5 mg suspension taken orally after surgery.
  Arms: V117957
Drug: Ibuprofen — Ibuprofen 400 mg tablets taken orally after surgery.
  Arms: Ibuprofen
Drug: Placebo — Placebo taken orally after surgery.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the analgesic properties of an oral dose of V117957 4.5 mg aqueous suspension in the third molar extraction model

ELIGIBILITY:
Inclusion Criteria include:

* Males aged 18 to 45 years;
* Females aged 18 to 45 years of nonchildbearing potential;
* A body mass index of 18 to 30.0 kg/m2, inclusive;
* Scheduled to undergo outpatient surgical extraction of 2 or more third molars (with at least 1 partial bony mandibular extraction);
* Experience moderate to severe pain;
* Use only topical benzocaine, 2% lidocaine with epinephrine, and nitrous oxide as preoperative medication;
* Are deemed by the investigator to be appropriate candidates for the protocol-specified therapeutic regimen.

Exclusion Criteria include:

* Are female who are pregnant, lactating or of child-bearing potential, or who have a positive pregnancy test result at screening or check-in;
* A history or any current conditions that might interfere with drug absorption, distribution, metabolism or excretion;
* A history of frequent nausea or emesis regardless of etiology;
* A history of seizures or head trauma with sequelae;
* A cardiovascular disorder, including hypertension, unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure or active myocardial ischemia;
* A history of alcohol or substance abuse or addiction;
* A history of opioid abuse or addiction;
* A positive urine drug or alcohol test at screening or check-in;
* A positive urine cotinine test result at screening or check-in, smokes frequently (>1 time per week) or have used tobacco or nicotine substitutes within 1 month before the loading dose of study drug, and/or have an inability to refrain from use of nicotine between check-in and the follow-up visit;
* Ingest xanthine- or caffeine-containing foods or beverages (eg, coffee, tea, chocolate, and colas) within 24 hours before the loading dose of study drug and for the duration of confinement to the clinical site;
* Have the presence or history (within 2 years of screening) of bleeding disorder(s) or peptic ulcer disease;
* Have donated or lost ≥ 500 mL of blood in the 60 days before screening;
* Use of any medication, other than those that are standard for dental surgery;
* Have used acetaminophen, ibuprofen, aspirin, or other nonsteroidal anti-inflammatory drugs or any other analgesics (OTC or prescription) within 3 days before surgery; or have used long-acting anesthetics (eg, bupivacaine) or any other medications that may result in prolonged anesthesia, analgesia, or sedation;
* Have presence of a chronic or acute painful condition, other than the study indication, which could interfere with the assessment of efficacy of the study drug or any other condition that, in the opinion of the investigator, would adversely affect the subject's ability to complete the study or its measures;
* Are unsuitable to participate in this study for any other reason, in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Total pain relief 0 to 8 hours after dosing (TOTPAR8) | 0 - 8 hours postdose
  Time-weighted sum of pain relief scores 0 to 8 hours after dosing

SECONDARY OUTCOMES:
Total Pain Relief 0 - 4 hours after dosing (TOTPAR4) | Hour 4 postdose
Total Pain Relief 0 - 6 hours after dosing (TOTPAR6) | Hour 6 postdose
Total Pain Relief 0 - 12 hours after dosing (TOTPAR12) | Hour 12 postdose
Total Pain Relief 0 - 24 hours after dosing (TOTPAR24) | Hour 24 postdose
Pain Relief (PR) over time | Up to 24 hours postdose
Pain intensity difference over time | 15, 30, 45 , 60, 90 minutes; 2, 3, 4, 4.5, 6, 8, 10, 12 and 24 hours postdose
Sum of pain intensity difference 0 to 4 hours after dosing (SPID4) | Hour 4 postdose
Sum of pain intensity difference 0 to 6 hours after dosing (SPID6) | Hour 6 postdose
Sum of pain intensity difference 0 to 8 hours after dosing (SPID8) | Hour 8 postdose
Sum of pain intensity difference 0 to 12 hours after dosing (SPID12) | Hour 12 postdose
Sum of pain intensity difference 0 to 24 hours after dosing (SPID24) | Hour 24 postdose
Time to first perceptible PR | Up to 24 hours postdose
Time to meaningful PR | Up to 24 hours postdose
Time to first use of rescue pain medication | Up to 24 hours postdose
Proportion of subjects taking rescue medication by time point | Up to 24 hours postdose
Global assessment of overall satisfaction | Hour 24 postdose

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Dental Pain Clinic, Austin, Texas, United States